CLINICAL TRIAL: NCT04369872
Title: Microwave Ablation of Primary and Secondary Lung Malignancies: A Phase I-II Single Centre Prospective Safety and Efficacy Trial
Brief Title: Microwave Ablation of Primary and Secondary Lung Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-19-0304
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-04

CONDITIONS: Lung Neoplasms; Neoplasm Metastasis
Keywords: Lung Cancer; Lung Metastases
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microwave Ablation (Experimental): Study participants will receive percutaneous microwave ablation of their malignant lung neoplasm.
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — Microwave ablation of lung lesion using Solero Microwave Tissue Ablation system.

SUMMARY:
Surgery is the first choice of treatment for early-stage primary pulmonary malignancies, but up to 15% of all patients, and 33% of patients greater than 75 years of age, are not surgical candidate's due to locally advanced disease, poor cardiopulmonary reserve and significant medical co-morbidities. Some patients are also unwilling to undergo surgery. This has prompted the development of alternatives to surgery so that local control of unresectable tumors can be achieved.

Stereotactic body radiation therapy (SBRT) is currently an alternative therapy for these patients with 3-year survival rates of between 42 and 60%. SBRT has excellent local control rates and a favorable toxicity profile relative to other surgical and non-surgical therapies. Radiation pneumonitis (RP), amongst others, is one of the major toxicities which can limit the maximal radiation dose that can be safely delivered to thoracic tumors. Reported rates of SBRT induced RP requiring clinical intervention range from 0% to 29% and life-threatening toxicities have been reported in up to 12% of cases in various studies. The potential for toxicities from SBRT could limit the number of times a patient could be treated with SBRT for residual, recurrent or new pulmonary lesions over time.

Following the first report of thermal ablation for lung malignancies in 2000, this modality has been used to treat primary and secondary malignancies and has emerged as an effective, low-cost, safe and repeatable alternative to SBRT for local tumour control. The most widely practised technique is radiofrequency ablation (RFA). Microwave ablation (MWA) is a relatively new therapy and offers all the advantages of RFA, but with significant additional advantages 3. These include reduced procedure times, lower complication rates, increased ablative temperatures, improved propagation of thermal energy particularly in the lung, improved efficacy in lesions that are in close proximity to blood vessels due to reduced heat-sink effect, and less procedure associated pain 2,3. Using high energy MWA to treat 87 pulmonary tumors, Egashira et al achieved a primary technical success rate of 94% and technique effectiveness of 98% at a median of 15 months.

MWA is performed by Interventional Radiologists using CT guidance. The treatment is performed under general anaesthesia and is repeatable. Multiple lesions can be ablated in one treatment session. Patients can potentially be discharged the same day of treatment, if there are no adverse events.

MWA is a relatively new treatment option that could be considered in situations where the patient is not a candidate for further treatment with surgery, SBRT or chemotherapy, or the patient declines the recommended standard available treatments.

Objectives for Phase I:

The primary objective for Phase I of this study will be to demonstrate the Safety of MWA performed for treatment of lung malignancy in patients not suitable for surgery, chemotherapy or SBRT.

Primary objective (Safety): to determine the proportion of patients experiencing local adverse events at one week definitively related to the mwa procedure.

Secondary objective (Feasibility): To determine the proportion of patients in whom technical success of MWA was achieved by assessing completion of ablation on CT at the time of the procedure, indicated by replacement of tumor by ground glass change (including a 5mm ablation zone in normal surrounding lung parenchyma).

Objectives for Phase II Primary objective (Efficacy): To demonstrate efficacy by measuring the proportion of patients demonstrating absence of residual tumor on follow up CT at 1 month after MWA.

Secondary objective: To determine the proportion of patients needing re-treatment for recurrent tumor at 1 month post MWA.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell Lung Carcinoma and metastatic lesions from lung, colorectal, breast, sarcoma, melanoma
* Patient median estimate survival of > 1 year, as determined by the treating physician
* ECOG 0-1
* <5 lesions in either lung
* Limited and/or controlled extra-pulmonary disease - to be determined by multidisciplinary consensus
* Not amenable to surgery, SBRT or chemotherapy (or patient refusal)
* Patient will have documentation by surgeon and/or radiation oncologist that the patient is unamenable to surgery and SBRT

Exclusion Criteria:

* Lesions >3cm in size
* Lesions within 1 cm of any critical mediastinal structure (e.g. aorta, main pulmonary arteries, esophagus, phrenic nerve), diaphragm or pleura
* FEV1≤35% predicted
* Clinically significant emphysema (to be determined by the treating physician)
* Previous pneumonectomy
* Inability to tolerate pneumothorax as judged by referring clinician's clinical assessment
* Inability to tolerate general anaesthetic
* Inability to provide informed consent
* INR > 1.5
* Platelets < 100
* PTT > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse outcomes following microwave ablation | 1 week post treatment
  Proportion of patients experiencing local adverse events at one week definitively related to the mwa procedure.
Efficacy of microwave ablation of lung lesions | 1 month post treatment
  To demonstrate efficacy by measuring the proportion of patients demonstrating absence of residual tumor on follow up CT at 1 month after MWA.
Rate of technical success | 1 month post treatment
  Proportion of patients in whom technical success of MWA was achieved by assessing completion of ablation on CT at the time of the procedure, indicated by replacement of tumor by ground glass change (including a 5mm ablation zone in normal surrounding lung parenchyma).

SECONDARY OUTCOMES:
Re-treatment rate. | 1 month post treatment
  To determine the proportion of patients needing re-treatment for recurrent tumor at 1 month post MWA.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Przybojewski, MB ChB, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberya, Canada

IPD SHARING:
Plan to Share IPD: No